CLINICAL TRIAL: NCT06569277
Title: Effects of a Smartphone Mobile Application on Quality of Bowel Preparation: A Randomized Controlled Trial
Brief Title: Impact of a Colonoscopy Preparation Mobile App on Colonoscopic Cleanliness and Experience
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital (Other)
Responsible Party: Principal Investigator, selim demirci, Clinical physician, Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: mobilapplication
Record Dates: First submitted 2024-08-22; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Bowel Preparation; Patient Experience; Patient Satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: All elective colonoscopies were performed by two experienced endoscopists who were unaware of the group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The mobile application group (Experimental): The research protocol was explained during the colonoscopy appointment, and patients, when they agreed to follow their diet to the mobile application, were accepted as part of the patient intervention group.
  Interventions: Other: A mobile application
- Control (No Intervention): The control group consists of patients who prepared for colonoscopy with the standard low-residue diet list.

INTERVENTIONS:
Other: A mobile application — Those who agreed to download a mobile app for colonoscopic bowel preparation on their smartphones.
  Arms: The mobile application group

SUMMARY:
The most crucial factor determining the success and quality of a colonoscopy procedure is the patient's adherence to proper bowel preparation. When a colonoscopy is scheduled, patients are provided with a diet plan designed to improve the quality of bowel cleansing, in addition to bowel-cleansing medications, through the endoscopy secretariat. Typically, in cases of inadequate bowel cleansing, where the bowel wall is not sufficiently visible during the colonoscopy, it is found that patients have poor adherence to the diet plan and have consumed incorrect or insufficient foods. This inadequate bowel cleansing can lead to missed pathologies such as polyps, colitis, diverticulosis, angiodysplasia, and cancer, which may cause patient complaints or symptoms.

Currently, patients who come to our secretariat from various clinics and polyclinics for colonoscopy appointments receive a single-page informational sheet containing a 5-day pre-procedure diet plan. In our study, the investigators aim to increase patient adherence to the colonoscopy diet by providing a comprehensive mobile application that includes recommendations and recipes for the foods listed in the colonoscopy preparation diet plan. This randomized study will involve selecting suitable patients who have accepted our study from routine colonoscopy requests and analyzing the impact of this mobile application on the quality of colon cleansing, the time to reach the cecum, and the detection rate of colon polyps.

The quality of bowel cleansing will be assessed using the Boston Bowel Preparation Score, where a score of 6 or higher for the entire colon and scores above 2 for each individual segment indicate adequate cleaning. The time to reach the cecum will be tracked using a stopwatch on our mobile phone during the colonoscopy, and the rate of colon polyp detection will be retrospectively reviewed after the study concludes.

The goal of this study is to enhance patient adherence through a free mobile application and to reduce unnecessary administrative costs.

DETAILED DESCRIPTION:
A total of 104 patients were included in this study. At the time of scheduling an outpatient colonoscopy, intervention group and control group were randomly assigned using a random-number generator for treatment allocation. The research protocol was explained during the colonoscopy appointment, and patients, when the participants agreed to follow their preparation to the mobile application, were accepted as part of the patient intervention group. A consent form was signed and collected. The nurse responsible for patient education in the endoscopy secretariat informed the patient that this mobile application is an important component of bowel preparation and adhere strictly to the recipes and recommendations. The group who received the standard diet list and applied for their colonoscopy appointments were randomly designated as the control group. Bowel preparation was evaluated during the colonoscopy using the Boston Bowel Preparation Scale (BBPS). Cecal insertion and withdrawal times, polyp detection rate, utilization of the recipe resource, and patients' experiences related to colonoscopy were recorded.

The research team utilized freely available resources from general cookery recipe websites to create the recipes, adapting it to align with the recommendations for a low-residue diet . Recipes were selected based on criteria such as being visually appealing, easy to prepare, and easily modifiable to comply with the low-residue diet. A dietitian examined the recipes to guarantee that the recipes followed low-residue diet guidelines. The colon preparation recommendations have been obtained from free medical information websites on the internet to facilitate adherence to bowel cleansing.

ELIGIBILITY:
Inclusion Criteria:

- All outpatients who apply for a colonoscopy appointment.

Exclusion Criteria:

* Patients with a history of prior colonoscopic procedures
* Using anticholinergic or gastrointestinal motility-reducing drugs
* Severe chronic kidney failure (GFR<30 ml/min)
* Advanced heart failure (NYHA III-IV)
* History of abdominal surgery were not included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2024-06-15 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Boston Bowel Preparation Scale (BBPS) | immediately after the procedure
  The BBPS is used to evaluate the quality of bowel preparation, with a scale from 0 to 9 (0 = very poor, 9 = excellent). Total BBPS score ≥ 6 and three segments of the colon (right, transverse, and the left side of the colon) ≥ 2 accepted as good bowel preparation

SECONDARY OUTCOMES:
cecal insertion time(minutes) | during the procedure
  Insertion time, as defined, refers to the duration between the initiation of the colonoscopy procedure and the moment when the endoscope reaches the cecum, with identification of the appendiceal orifice.
withdrawal time (minutes) | during the procedure
  Withdrawal time, as defined, refers to the period between the commencement of withdrawing the colonoscope from the cecum and the complete removal of the colonoscope from the patient.
polyp detection rate | during the procedure
  It will be assessed by recording the encountered polyps during colonoscopy.
patient experience | immediately after the procedure
  The patient experience of the study group was evaluated using a 3-point scale (1-worse than expected, 2-as expected, 3-better than expected).

CONTACTS AND LOCATIONS:
Overall Officials: selim demirci, Principal Investigator — clinical physician
Locations (1):
- Abdurrahman Yurtaslan Oncology and Training Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zhao K, Dong R, Xia S, Feng L, Zhou W, Zhang M, Zhang Y, Tian D, Liu M, Liao J. Improving the quality of bowel preparation by smartphone education platform prior to colonoscopy: a randomized trail. Ann Med. 2022 Dec;54(1):2777-2784. doi: 10.1080/07853890.2022.2130972. PMID 36254495
- [Result] Dao HV, Dao QV, Lam HN, Hoang LB, Nguyen VT, Nguyen TT, Vu DQ, Pokorny CS, Nguyen HL, Allison J, Goldberg RJ, Dao ATM, Do TTT, Dao LV. Effectiveness of using a patient education mobile application to improve the quality of bowel preparation: a randomised controlled trial. BMJ Open Gastroenterol. 2023 Jun;10(1):e001107. doi: 10.1136/bmjgast-2023-001107. PMID 37277203
- [Result] van der Zander QEW, Reumkens A, van de Valk B, Winkens B, Masclee AAM, de Ridder RJJ. Effects of a Personalized Smartphone App on Bowel Preparation Quality: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2021 Aug 19;9(8):e26703. doi: 10.2196/26703. PMID 34420924
- [Derived] Demirci S, Sezer S. Effects of a smartphone mobile application on quality of bowel preparation: A randomized controlled trial. Pak J Med Sci. 2025 Jul;41(7):1905-1912. doi: 10.12669/pjms.41.7.11852. PMID 40735592